CLINICAL TRIAL: NCT00995683
Title: Effect of Preventive Sodium Lactate Infusion on Intracranial Hypertension in Severe Trauma Tic Brain Injury
Brief Title: Preventive Sodium Lactate and Traumatic Brain Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Collaborators: Université de Nice Sophia Antipolis (Other); Medical University of Grenoble (Other)
Responsible Party: Carole Ichai, Institut d'Anesthésiologie des Alpes Maritimes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PA-Lac-TBI
Record Dates: First submitted 2009-10-10; First posted 2009-10-15 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-05

CONDITIONS: Head Trauma
Keywords: intracranial hypertension; neurological outcome; osmotherapy
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hypertension | interventions — Sodium Lactate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- half sodium lactate (Experimental): infusion of 0.5 ml/kg/day during 48 hours
  Interventions: Drug: half molar sodium lactate
- isotonic sodium chloride (Active Comparator): infusion of 0.5 ml/kg during 48 hours
  Interventions: Drug: isotonic sodium chloride

INTERVENTIONS:
Drug: half molar sodium lactate — intravenous infusion of 0.5 ml/kg during 48 hours
  Other Names: sodium lactate
  Arms: half sodium lactate
Drug: isotonic sodium chloride — intravenous infusion of 0.5 ml/kg during 48 hours
  Other Names: sodium chloride
  Arms: isotonic sodium chloride

SUMMARY:
The goal of this study is to evaluate the effect of preventive intravenous infusion of half molar sodium lactate on the onset of hypertensive intracranial episodes in severe head trauma. The investigators hypothesize that preventive intravenous administration of sodium lactate will decrease the number of treatments required to decrease intracranial pressure during 48 hours.

DETAILED DESCRIPTION:
* Intracranial hypertension is the most severe complication of severe head injury. This may lead to cerebral death or severe neurological outcome. To improve the prognosis of these patients,intracranial pressure must be maintained in normal range while maintaining cerebral perfusion pressure. Among numerous strategies, osmotherapy is frequently proposed to decrease intracranial pressure, using mannitol or hypertonic saline. Recently, it has been found that hypertonic sodium lactate infusion is more efficient to decrease intracranial hypertension compared with an equivalent volemic and osmotic mannitol administration.Thus, we hypothesized that a preventive sodium lactate infusion in severe head trauma could decrease the number of intracranial hypertensive episodes.
* Methods and Objectives : to compare in a randomized double-blind fashion two group of patients, i.e., those receiving a standard isotonic saline infusion (control group) with those receiving half-molar sodium lactate for 48 hours following admission in ICU. The primary endpoint is the number of any treatment required to control intracranial hypertensive episodes occurring during the first 48 hours following admission in ICU. Secondary endpoints are the effect of sodium lactate infusion on : intracranial pressure evolution;neurological outcome at 6 months (glasgow outcome scale); cerebral blood flow evaluated by transcranial doppler; and daily water balance
* Protocol consisted to measure as soon as possible baseline intracranial pressure and cerebral perfusion pressure, then immediately to begin the administration of 0.5 ml/kg/h intravenous isotonic saline perfusion or half-molar sodium lactate during 48 hours in a randomized double-blind fashion. Management of patients is the same for all patients. Treatment required for intracranial hypertensive episode is decided by a senior physician in charge of the patient. Sample size has been calculated considering that 50% of these patients will develop at least one intracranial hypertensive episode, each of them requiring at least 2 treatments. Based on previous results, we hypothesized that sodium lactate will decrease the number of required treatment by 2, leading to a sample size of 30 patients per group
* Follow up : 48 hours for treatments of intracranial hypertensive episodes; 6 months for the neurological outcome (glasgow outcome scale)

ELIGIBILITY:
Inclusion Criteria:

* severe head trauma with a glasgow coma scale less than 9

Exclusion Criteria:

* prehospital cardiac arrest
* severe hemorrhage shock
* severe circulatory or respiratory failure
* medullar trauma
* prehospital osmotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
the number of treatments required for intracranial hypertensive episodes during the first 48 hours following ICU admission | 48 hours

SECONDARY OUTCOMES:
the neurological outcome at six months evaluated by the glasgow outcome scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ichai, MD, PhD, Principal Investigator — Institut d'Anesthesiologie des Alpes Maritimes
Locations (1):
- Institut d'Anesthesiologie des Alpes maritimes, Nice, Nice, France

REFERENCES:
- [Result] Ichai C, Armando G, Orban JC, Berthier F, Rami L, Samat-Long C, Grimaud D, Leverve X. Sodium lactate versus mannitol in the treatment of intracranial hypertensive episodes in severe traumatic brain-injured patients. Intensive Care Med. 2009 Mar;35(3):471-9. doi: 10.1007/s00134-008-1283-5. Epub 2008 Sep 20. PMID 18807008